CLINICAL TRIAL: NCT01464177
Title: Prospective Randomized Phase II Trial of Hypofractionated Stereotactic Radiotherapy in Recurrent Glioblastoma Multiforme
Brief Title: Hypofractionated Stereotactic Radiotherapy in Recurrent Glioblastoma Multiforme
Acronym: GBM Hypo RT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Andre Tsin Chih Chen (Other)
Responsible Party: Sponsor-Investigator, Andre Tsin Chih Chen, Medical Doctor, University of Sao Paulo
Organization: University of Sao Paulo (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RT-01/2011
Record Dates: First submitted 2011-10-25; First posted 2011-11-03 (Estimated); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Recurrent Glioblastoma Multiforme
Keywords: malignant glioma; glioblastoma; radiotherapy; randomized
MeSH Terms: conditions — Glioblastoma; Glioma

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Stereotactic hypofractionated RT 5x5Gy (Active Comparator): Stereotactic hypofractionated radiation therapy delivered as follows:
  * Gross tumor volume (GTV) equals enhancement area in T1 contrast enhanced MRI.
  * Planning tumor volume (PTV) equals GTV plus 3mm margin.
  * the dose of radiation will be 25Gy delivered in 5 fractions.1 fraction per day, non consecutive days in a maximum period of 10 working days.
  * RT to begin in a maximum of 2 weeks after randomization.
  Interventions: Radiation: Stereotactic hypofractionated RT 5x5Gy
- Stereotactic hypofractionated RT 5x7Gy (Experimental): Stereotactic hypofractionated radiation therapy delivered as follows:
  * Gross tumor volume (GTV) equals enhancement area in T1 contrast enhanced MRI.
  * Planning tumor volume (PTV) equals GTV plus 3mm margin.
  * the dose of radiation will be 35Gy delivered in 5 fractions.1 fraction per day, non consecutive days in a maximum period of 10 working days.
  * RT to begin in a maximum of 2 weeks after randomization.
  Interventions: Radiation: Stereotactic hypofractionated RT 5x7Gy

INTERVENTIONS:
Radiation: Stereotactic hypofractionated RT 5x5Gy — Stereotactic hypofractionated radiation therapy delivered as follows:
  * Gross tumor volume (GTV) equals enhancement area in T1 contrast enhanced MRI.
  * Planning tumor volume (PTV) equals GTV plus 3mm margin.
  * The dose of radiation will be 25Gy delivered in 5 fractions.1 fraction per day, non consecutive days in a maximum period of 10 working days.
  * RT to begin in a maximum of 2 weeks after randomization
  Arms: Stereotactic hypofractionated RT 5x5Gy
Radiation: Stereotactic hypofractionated RT 5x7Gy — Stereotactic hypofractionated radiation therapy delivered as follows:
  * Gross tumor volume (GTV) equals enhancement area in T1 contrast enhanced MRI.
  * Planning tumor volume (PTV) equals GTV plus 3mm margin.
  * The dose of radiation will be 35Gy delivered in 5 fractions.1 fraction per day, non consecutive days in a maximum period of 10 working days.
  * RT to begin in a maximum of 2 weeks after randomization.
  Arms: Stereotactic hypofractionated RT 5x7Gy

SUMMARY:
Glioblastoma multiforme (GBM) is the most common primary brain tumor in adults. The treatment comprises maximal safe resection followed by radiotherapy and chemotherapy. Despite appropriate management, 90% of the patients will develop relapse or progression. After progression, the median survival is 5.2 months (Stupp, 2009).

The treatment of GBM relapse remains investigational. Reirradiation is an option in selected cases.

The objective of this study is to compare 2 schemes of stereotactic hypofractionated radiotherapy in the management of recurrent GBM.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* KPS equal or greater than 60
* Anatomopathological confirmation of GBM
* Previous RT with therapeutic doses
* At least 5 months from the end of RT course
* Not a candidate to surgical resection
* Patients with partial resection after resection of recurrent GBM will be allowed
* Patients with local progression after resection of recurrent GBM will be allowed
* Lesion with a maximal 150cc volume, as defined by enhancing portion in contrast enhanced MRI
* Hemoglobin levels (Hb) equal or greater than 10ng/dl. Blood transfusions to correct the Hb will be allowed.

Exclusion Criteria:

* Important comorbidities
* Concomitant chemotherapy
* Contraindication to MRI
* Brainstem glioma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2011-10 (Actual); Primary Completion 2021-07 (Actual); Study Completion 2024-08 (Actual)

PRIMARY OUTCOMES:
progression free survival | from date of randomization until date of first documented progression or death from any cause, which ever comes first, assessed up to 48 months
  progression free survival as defined by the "Response Assesment in Neuro Oncology Working Group"(Wen, 2010). Briefly progression is defined as:
  * increase in 25% of the product of perpendicular diameters of enhancing lesions
  * significant increase in T2/Flair non enhancing component
  * appearance of new lesions
  * clinical deterioration not attributable to other causes other than the tumor or reduction in corticosteroid dose

SECONDARY OUTCOMES:
overall survival | from date of randomization until death from any cause, assessed up to 48 months
local control | from date of randomization until date of local progression, assessed up to 48 months
toxicity | from date of randomization until death, assessed up to 48 months
  * toxicity scored by the Common Terminology of Adverse Events version 4
  * will be assessed every 2 months or in case of patient hospitalization or visit to the E.R.
quality of life | from date of randomization until last follow-up, assessed up to a period of 48 months
  * quality of life measured by the "FACT Br" questionary
  * will be assessed every 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Andre T Chen, M.D. / PhD, Principal Investigator — Hospital das Clinicas da Faculdade de Medicina da USP
Locations (1):
- Hospital das Clinicas da Faculdade de Medicina da USP, São Paulo, São Paulo, Brazil

REFERENCES:
- [Background] Stupp R, Mason WP, van den Bent MJ, Weller M, Fisher B, Taphoorn MJ, Belanger K, Brandes AA, Marosi C, Bogdahn U, Curschmann J, Janzer RC, Ludwin SK, Gorlia T, Allgeier A, Lacombe D, Cairncross JG, Eisenhauer E, Mirimanoff RO; European Organisation for Research and Treatment of Cancer Brain Tumor and Radiotherapy Groups; National Cancer Institute of Canada Clinical Trials Group. Radiotherapy plus concomitant and adjuvant temozolomide for glioblastoma. N Engl J Med. 2005 Mar 10;352(10):987-96. doi: 10.1056/NEJMoa043330. PMID 15758009
- [Background] Stupp R, Hegi ME, Mason WP, van den Bent MJ, Taphoorn MJ, Janzer RC, Ludwin SK, Allgeier A, Fisher B, Belanger K, Hau P, Brandes AA, Gijtenbeek J, Marosi C, Vecht CJ, Mokhtari K, Wesseling P, Villa S, Eisenhauer E, Gorlia T, Weller M, Lacombe D, Cairncross JG, Mirimanoff RO; European Organisation for Research and Treatment of Cancer Brain Tumour and Radiation Oncology Groups; National Cancer Institute of Canada Clinical Trials Group. Effects of radiotherapy with concomitant and adjuvant temozolomide versus radiotherapy alone on survival in glioblastoma in a randomised phase III study: 5-year analysis of the EORTC-NCIC trial. Lancet Oncol. 2009 May;10(5):459-66. doi: 10.1016/S1470-2045(09)70025-7. Epub 2009 Mar 9. PMID 19269895
- [Background] Niyazi M, Siefert A, Schwarz SB, Ganswindt U, Kreth FW, Tonn JC, Belka C. Therapeutic options for recurrent malignant glioma. Radiother Oncol. 2011 Jan;98(1):1-14. doi: 10.1016/j.radonc.2010.11.006. Epub 2010 Dec 13. PMID 21159396
- [Background] Shepherd SF, Laing RW, Cosgrove VP, Warrington AP, Hines F, Ashley SE, Brada M. Hypofractionated stereotactic radiotherapy in the management of recurrent glioma. Int J Radiat Oncol Biol Phys. 1997 Jan 15;37(2):393-8. doi: 10.1016/s0360-3016(96)00455-5. PMID 9069312
- [Background] Vordermark D, Kolbl O, Ruprecht K, Vince GH, Bratengeier K, Flentje M. Hypofractionated stereotactic re-irradiation: treatment option in recurrent malignant glioma. BMC Cancer. 2005 May 30;5:55. doi: 10.1186/1471-2407-5-55. PMID 15924621
- [Background] Ernst-Stecken A, Ganslandt O, Lambrecht U, Sauer R, Grabenbauer G. Survival and quality of life after hypofractionated stereotactic radiotherapy for recurrent malignant glioma. J Neurooncol. 2007 Feb;81(3):287-94. doi: 10.1007/s11060-006-9231-0. Epub 2006 Sep 20. PMID 17031558
- [Background] Fogh SE, Andrews DW, Glass J, Curran W, Glass C, Champ C, Evans JJ, Hyslop T, Pequignot E, Downes B, Comber E, Maltenfort M, Dicker AP, Werner-Wasik M. Hypofractionated stereotactic radiation therapy: an effective therapy for recurrent high-grade gliomas. J Clin Oncol. 2010 Jun 20;28(18):3048-53. doi: 10.1200/JCO.2009.25.6941. Epub 2010 May 17. PMID 20479391
- [Background] Fokas E, Wacker U, Gross MW, Henzel M, Encheva E, Engenhart-Cabillic R. Hypofractionated stereotactic reirradiation of recurrent glioblastomas : a beneficial treatment option after high-dose radiotherapy? Strahlenther Onkol. 2009 Apr;185(4):235-40. doi: 10.1007/s00066-009-1753-x. Epub 2009 Apr 16. PMID 19370426
- [Background] Cheng JX, Zhang X, Liu BL. Health-related quality of life in patients with high-grade glioma. Neuro Oncol. 2009 Feb;11(1):41-50. doi: 10.1215/15228517-2008-050. Epub 2008 Jul 15. PMID 18628405
- [Background] Liu R, Page M, Solheim K, Fox S, Chang SM. Quality of life in adults with brain tumors: current knowledge and future directions. Neuro Oncol. 2009 Jun;11(3):330-9. doi: 10.1215/15228517-2008-093. Epub 2008 Nov 10. PMID 19001097
- [Background] Wen PY, Macdonald DR, Reardon DA, Cloughesy TF, Sorensen AG, Galanis E, Degroot J, Wick W, Gilbert MR, Lassman AB, Tsien C, Mikkelsen T, Wong ET, Chamberlain MC, Stupp R, Lamborn KR, Vogelbaum MA, van den Bent MJ, Chang SM. Updated response assessment criteria for high-grade gliomas: response assessment in neuro-oncology working group. J Clin Oncol. 2010 Apr 10;28(11):1963-72. doi: 10.1200/JCO.2009.26.3541. Epub 2010 Mar 15. PMID 20231676